CLINICAL TRIAL: NCT01821690
Title: Brain Research in Aggression and Irritability Network (BRAIN): Building Evidence-Based Approaches to Managing Traumatic Brain Injury
Brief Title: Buspirone for the Treatment of Traumatic Brain Injury (TBI) Irritability and Aggression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Flora Hammond, Covalt Professor and Chair, Physical Medicine and Rehabilitation, Indiana University School of Medicine Chief of Medical Affairs, Rehabilitation Hospital of Indiana, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1210009885; CFDA #: 84.133A-120035 (Other Grant/Funding Number: National Institute on Disability and Rehabilitation Research)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Buspirone; Behavior; Irritability; Aggression
MeSH Terms: conditions — Brain Injuries, Traumatic; Behavior; Aggression | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buspirone Treatment (Experimental): starting at 15 mg/day and ending at 60 mg/day as prescribed
  Interventions: Drug: Buspirone
- Buspirone Placebo (Placebo Comparator): placebo tablets as prescribed
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Buspirone/placebo will be given in increasing increments of 15 mg as needed. Subjects will start with 15 mg on day one and end with 60 mg on day 91 or placebo equivalent. Dose is titrated based on treatment response.
  Other Names: Buspar
  Arms: Buspirone Treatment
Drug: Placebo — The placebo tablets taste and look identical to buspirone.
  Arms: Buspirone Placebo

SUMMARY:
The purpose of this study is to improve behavior control displayed by persons with traumatic brain injury by assessing effectiveness of treatments for post-TBI irritability and aggression.

DETAILED DESCRIPTION:
PURPOSE OF PROJECT: To study the effect expressed by persons with TBI through assessment of buspirone effectiveness for post-traumatic irritability and aggression and development of an irritability/aggression impact measure.

SUMMARY OF PROJECT: It is anticipated that 74 subjects with 74 corresponding subject observers will be recruited for the treatment study. Subjects will be recruited from community and self-referrals.

Interested potential participants will be scheduled for an in-person screening visit. Subjects who consent and qualify will be randomized in a 1:1 ratio, buspirone or placebo. Stratification to randomization group will occur based on the presence of major or minor depression (defined by PHQ-9 total score >5). Randomized subjects will receive active treatment or placebo. There will be 4 clinic visits. Visits will occur at baseline, for consenting and screening, day 35, day 63 and day 91. At all 4 clinic visits, both the subject and the observer will be given questionnaires regarding the subject's behavior and mood. Day 91 ends the period of the randomized clinical trial phase of the study and the subjects will begin the 1 month continuation phase of the study in which all participants receive active buspirone.

The following questionnaires will be used as measures of irritability and aggression for the subject and the observer: Neuropsychiatric Inventory (NPI & NPI-Distress), Aggression & Irritability Impact Measure (AIIM) and Global Impression of Change.

The following questionnaires will be dispensed to the subject only: TBI-Quality of Life-Anger, Personal Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), PTSD Checklist Civilian (PCL-C), and Glasgow Outcome Scale Extended (GOS-E) The Investigator will complete the Clinical Global Impression of change at Visits 1, 2, 3, and 4. History and Physical Exam, creatinine level (kidney function) and liver function tests will be obtained for eligibility. Serum pregnancy tests will be drawn at screening for females of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Closed head injury (impaired brain function resulting from externally inflicted trauma without penetrating injury as defined below) at least 6 months prior to enrollment
* Irritability that is either new or worse than level of irritability before the traumatic brain injury, by report of observer or person with TBI
* Age at time of enrollment: 18 to 70 years
* Voluntary informed consent of patient and observer
* Subject and observer willing to comply with the protocol
* Observer-rated NPI Irritability Domain score 6 or greater to include only moderate-severe irritability
* Medically and neurologically stable during the month prior to enrollment.
* If taking antidepressant, anxiolytic, hypnotic, or stimulant medications, no change anticipated in these medications during the month prior to enrollment
* No change in therapies or medications planned during the 91-day participation
* No surgeries planned during the 91-day participation
* Vision, hearing, speech, motor function, and comprehension sufficient for compliance with all testing procedures and assessments
* Observer (e.g.: family member, close friend, employer) with whom subject interacts sufficiently to observe occurrences of irritability. The observer interacts with the participant for a period long enough and of a nature to be able to judge the participant's irritability. The interactions would need to be adequate to judge observer distress over the irritability, severity of irritability and frequency of irritability on the following scale: < once weekly; once per week; several times per week, but not every day; essentially continuous.

Exclusion Criteria:

* Potential subject without a reliable observer
* Penetrating head injury as defined by head injury due to gunshot, projectile or foreign object
* Injury < 6 months prior to enrollment
* Ingestion of buspirone during the month prior to enrollment
* Inability to interact sufficiently for communication with caregiver
* History of schizophrenia or psychosis
* Diagnosis of progressive or additional neurologic disease
* Clinical signs of active infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory-Irritability Domain | Day 91
  A self-report measure of irritability

SECONDARY OUTCOMES:
Neuropsychiatric Inventory-Aggression Domain | Day 91
  A self-report measure of aggression
Neuropsychiatric Inventory-Distress Irritability Domain | Day 91
  A self-report measure of the distress caused by irritability
Neuropsychiatric Inventory-Distress Aggression Domain | Day 91
  A self-report measure of the distress caused by aggression
St. Andrews-Swansea Neurobehavioural Outcome Scale | Day 91
  A self-report measure of overall neurobehavioral function
Personal Health Questionnaire | Day 91
  A measure of depression that maps on to DSM criteria for depression
Traumatic Brain Injury-Quality of Life Anger | Day 91
  A self-report measure of overall impact of anger on quality of life
Global Impressions of Change | Day 91
  A self-report measure of overall change
Clinical Global Impressions | Day 91
  Clinician rating of overall change
Aggression and Irritability Impact Measure | 91 Day
  A self-report measure of overall impact of irritability on life participation
Generalized Anxiety Disorder | 91 day
  A self-report measure of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Flora Hammond, MD, Principal Investigator — Indiana University/Rehabilitation Hospital of Indiana
Locations (1):
- Indiana University and Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be available upon request 24 months after completion of the project. Data requests should be submitted to the principal investigator.

REFERENCES:
- See also: Rehabilitation Hospital of Indiana — http://rhin.com
- See also: Indiana University School of Medicine — http://medicine.iu.edu